CLINICAL TRIAL: NCT06832150
Title: SMS 2: Impact of Cancer Therapy on the Somatic Mutational Landscape of Normal Tissues
Acronym: SMS2
Status: Enrolling by invitation | Type: Observational
Sponsor: The Wellcome Sanger Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 341204
Record Dates: First submitted 2025-02-05; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-07

CONDITIONS: Somatic Mutation; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, urine samples and cheek swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non melanoma skin cancer: Skin cancer patients receiving Immune checkpoint immunotherapy.
  Interventions: Other: sample collection; Other: Discussing study; Other: Seeking consent
- Head and Neck Cancer: Head and Neck cancer patients receiving chemoradiotherapy.
  Interventions: Other: sample collection; Other: Discussing study; Other: Seeking consent

INTERVENTIONS:
Other: sample collection — Participants may collected their own cheek swabs and will collect their own urine samples.
  Clinical professionals at participating sites will collect blood samples.
Other: Discussing study — Research Nurse/ Suitably qualified Research Site Staff will discuss the study with potential participants
Other: Seeking consent — Potential participants who wish to give consent will do with a Research Nurse/ Suitably qualified Research Site Staff.

SUMMARY:
Recently technology has been developed at the Wellcome Sanger Institute to allow clusters of cells with mutations to be detected in normal and diseased tissues. The researchers wish to determine how the number and nature of these mutant cell clusters change in response to treatments given to cancer patients (such as chemotherapy, radiotherapy, immunotherapy, and drugs targeted at specific mutations in tumours). As such the researchers wish to collect research samples of blood, cheek cells (via swabs) and urine from adult cancer patients receiving the above-mentioned treatments as part of their standard care. The researchers also wish to access any leftover tissue following surgery that is undertaken as part of these patient's treatment.

DETAILED DESCRIPTION:
Disease and tissue aging are thought to be influenced by genetic changes, or mutations, acquired throughout life. These mutations provide clues regarding the genetic damage that occurred through the lifetime of the patient, and include mutations caused by environmental factors such as ultraviolet light from sunlight or tobacco smoke affecting the skin or internal tissues, respectively. Other mutations may occur due to errors in copying the genome as cells divide. Once a cell has acquired a mutation, the cell's daughters may inherit it. Eventually clusters of cells carrying the same mutation may form within tissues. If the mutations alter cell behaviour this may impact how cells behave and influence how a whole tissue functions.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Due to commence systemic treatment for histologically confirmed cancer at a - participating site
* Age over 18 years
* Able to give informed consent.
* Able to give urine, blood and cheek swab samples on two occasions.
* Likely to complete 3 months of treatment

Exclusion Criteria:

* Anyone outside of the inclusion criteria plus individuals who Lack the capacity to provide informed consent and those who do not have a good command of the English language.
* Any participant who is known to have Hep B, Hep C or HIV

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is looking at two groups of patients having different types of cancer treatment in the study. A research nurse or clinician will highlight a potential participant for recruitment who is under their care and about to receive treatment for cancer. This will usually take place at the multidisciplinary team meeting.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2028-05-14 (Estimated); Study Completion 2029-05-13 (Estimated)

PRIMARY OUTCOMES:
To measure the frequency of acquired (somatic) mutations | 5 years
  The study will measure the frequency, size and nature of acquired (somatic) mutations in clusters of cells in normal blood, urinary tract and oral cells changes after cancer treatment.
To measure the size of acquired (somatic) mutations | 5 years
  The study will measure the size of acquired (somatic) mutations in clusters of cells in normal blood, urinary tract and oral cells changes after cancer treatment.

SECONDARY OUTCOMES:
To understand the nature of acquired (somatic) mutations | 5 years
  The study will attempt to define and/or understand the behaviour/ nature of acquired (somatic) mutations in clusters of cells in normal blood, urinary tract and oral cells changes after cancer treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Phil Jones, Principal Investigator — Wellcome Sanger Institute
Locations (1):
- Wellcome Sanger Institute, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No